CLINICAL TRIAL: NCT06525597
Title: A Randomized, Double-blind, Placebo-controlled Phase II Clinical Study Evaluating the Efficacy and Safety of Stapokibart Injection in Patients With Allergic Rhinitis
Brief Title: Study of Stapokibart Injection in Patients With Allergic Rhinitis
Acronym: MIZAR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM310-107101
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-08

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stapokibart Group (Experimental): Stapokibart, subcutaneous, once every two weeks
  Interventions: Biological: Stapokibart Injection
- Placebo Group (Placebo Comparator): Placebo, subcutaneous, once every two weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Stapokibart Injection — IL-4Rα monoclonal antibody
  Arms: Stapokibart Group
Drug: Placebo — Placebo
  Arms: Placebo Group

SUMMARY:
This study is a Randomized, Double-blind, Placebo-controlled phase II clinical study evaluating the efficacy and safety of Stapokibart injection in patients with allergic rhinitis.

DETAILED DESCRIPTION:
Allergic rhinitis (AR) is a non infectious chronic inflammatory disease of the nasal mucosa that is mainly mediated by immunoglobulin E (IgE) in atopic individuals exposed to allergens.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand the study and voluntarily sign the Informed consent form.
* Diagnosed Allergic Rhinitis according to the Criteria stated in the Chinese Guidelines for the Diagnosis and Treatment of Allergic Rhinitis (2022, Revised Edition).
* Subjects with asthma must be evaluated by the researcher as having a stable condition.
* Has a positive skin prick test (SPT) or positive antigen-specific serum immunoglobulin E (IgE).

Exclusion Criteria:

* Use of anti-interleukin 4 receptor alpha subunit (IL-4Rα) monoclonal antibody, thymic stromal lymphopoietin (TSLP) monoclonal antibody, anti-IgE monoclonal antibody, other monoclonal antibodies, or other biologics within 10 weeks or 5 half-lives (whichever is longer) prior to the screening visit.
* Use of any investigational product within 4 weeks prior to the screening visit or planning to participate in other clinical studies during this study.
* Forced expiratory volume in 1 second (FEV1) ≤ 50% of the predicted value during the screening/run-in period.
* Have acute sinusitis, nasal infection, or upper respiratory tract infection at screening or within 2 weeks prior to screening.
* Have received a live-attenuated vaccine within 12 weeks prior to randomization or planning to receive one during the study.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in daily reflective total nasal symptom scores (rTNSS) over 4 weeks of treatment. | Up to week 4
  The total nasal symptom score (TNSS) is the sum of the four symptom scores for rhinorrhea, nasal congestion, nasal itching, and sneezing, where each symptom is scored on a scale of 0 to 3.

CONTACTS AND LOCATIONS:
Overall Officials: Luo Zhang, Principal Investigator — Beijing Tong-Ren hospital
Locations (1):
- Beijing Tongren Hospital, CMU, Beijing, Beijing Municipality, China